CLINICAL TRIAL: NCT04622631
Title: the Use of 18F-FDG, 18F-DOPA and 68Ga-DOTATATE PET/CT in Patients With NETs That Are Potential Candidates for PRRT
Brief Title: Using 18F- FDG,18F-DOPA and 68Ga-DOTATATE PET/CT in Detection and Evaluation of Response in Patients With NET Undergoing PRRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Nayruz Knaana (Other Government)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Nayruz Knaana, Dr., Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-20- 6260-NK-CTIL
Record Dates: First submitted 2020-10-30; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Neuroendocrine Tumors
Keywords: Peptide Receptor Radionuclide treatment
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- PRRT positive: patients who have good response to prrt treatment - the tumor and/or the metastatic disease show no uptake/activity on PET-CT scans
- PRRT negative: no response to PRRT treatment

SUMMARY:
the investigators will follow up after patients with neuroendocrine tumors who undergo PRRT treatment and evaluate the response for treatment using PET/CT with different tracers

DETAILED DESCRIPTION:
patients with suspected or biopsy proven NET will undergo imaging using a Combination of 18F- FDG , 18F-DOPA and 68Ga-DOTATATE PET/CT before the stat of PRRT . after two cycles of treatment another two PET/CT are done using 18F- FDG and 18F-DOPA and about 6-8 weeks from last treatment the patient will undergo PET/CT using 18F-DOPA .

ELIGIBILITY:
Inclusion Criteria:

* patient with neuroendocrine tumor
* eligible for PRRT

Exclusion Criteria:

* younger than 18 years old
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with neuroendocrine tumor who were found to be eligible for Peptide Receptor Radionuclide Therapy (PRRT)
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with good response to Peptide Receptor Radionuclide Therapy (PRRT) | 7 months
  patients who have clinical and radiological improvement (using RECIST CRITERIA )
Number of participants with no response to Peptide Receptor Radionuclide Therapy (PRRT) treatment | 7 months
  patients who have no clinical and radiological improvement or worsening in clinical condition or radiologic findings (RECIST )

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel